CLINICAL TRIAL: NCT01093027
Title: Electrophysiological Study of the Effects of Limb Cooling on Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Virgilio Evidente, MD, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 09-007889
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Tremor
Keywords: Essential Tremor; Cooling; Temperature; Patients with Essential Tremor involving the upper limbs with at least moderate tremor.
MeSH Terms: conditions — Tremor; Essential Tremor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 15 - 30 (Other): The upper limb with tremor will be cooled with 15 degrees Celsius water for 10 minutes at Visit 1 and with 30 degrees Celsius water for 10 minutes at Visit 2.
  Interventions: Other: 15 - 30
- 30 - 15 (Other): The upper limb with tremor will be cooled with 30 degrees Celsius water for 10 minutes at Visit 1 and with 15 degrees Celsius water for 10 minutes at Visit 2.
  Interventions: Other: 30 - 15

INTERVENTIONS:
Other: 15 - 30 — The upper limb with tremor will be cooled with 15 degrees Celsius water for 10 minutes at Visit 1 and with 30 degrees Celsius water for 10 minutes at Visit 2.
  Arms: 15 - 30
Other: 30 - 15 — The upper limb with tremor will be cooled with 30 degrees Celsius water for 10 minutes at Visit 1 and with 15 degrees Celsius water for 10 minutes at Visit 2.
  Arms: 30 - 15

SUMMARY:
To determine the effects of upper limb forearm cooling on Essential Tremor upper limb tremor using a more practical method of limb cooling through a forearm cold pack.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of E.T. for at least a year by a movement disorder neurologist
* A +2 or worse action or kinetic tremor of one or both upper limbs involving at least the forearm and/or hand
* Ages 18 to 95 years old

Exclusion Criteria:

* (+) sensory loss in the upper extremities
* dermatologic lesions in upper extremities (e.g. skin cancer, eczema, fresh or healing wounds, abrasions, acne, pustules, abscesses, or skin rash)
* known history of sensitivity to cold (i.e., cold urticaria)
* known peripheral vascular disease
* Raynaud's phenomenon
* scleroderma

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virgilio Evidente, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Visits were scheduled between June 2010 and December 2011.
Period: Visit 1
Arm/Group | 15 - 30 | 30 - 15
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Visit 2
Arm/Group | 15 - 30 | 30 - 15
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 - 30 | 30 - 15 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 71.2 (6.8) | 76.3 (4.9) | 73.8 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Tremor Amplitude
Description: Average tremor amplitude during the Outstretched, Abducted, Nose, and Mug conditions of the Tremor Rating Scale test.
Time Frame: After 10 minutes of limb cooling treatment.
Measure: Mean (Standard Deviation); unit: cm/s^2
Arm/Group | 15 - 30 | 30 - 15
Number analyzed (Participants) | 10 | 10
cm/s^2
  Visit 1 | 127 (50) | 104 (44)
  Visit 2 | 150 (73) | 100 (58)

2. Secondary Outcome: Tremor Rating Scale
Description: Arm tremor severity was rated on a scale from 0=None to 4=Severe during each of four conditions: arm outstretched, hand close to mouth and arm abducted, performing a finger to nose maneuver, and holding a mug. The Tremor Rating Scale score was the mean of the scores for the four conditions, and ranged from a score of 0=None to 4=Severe.
Time Frame: After 10 minutes of limb cooling treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 15 - 30 | 30 - 15
Number analyzed (Participants) | 10 | 10
units on a scale
  Visit 1 | 1.35 (0.61) | 1.65 (0.49)
  Visit 2 | 1.68 (0.65) | 1.32 (0.47)

ADVERSE EVENTS:
Arm/Group | 15 - 30 | 30 - 15
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes